CLINICAL TRIAL: NCT00005092
Title: A Phase I Study of Photochemically Treated Donor T-Cell Supplements in HLA Haplotype Mismatched Hematopoietic Stem Cell Transplantation
Brief Title: Chemotherapy, Radiation Therapy, and Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-283; P30CA016672 (NIH); MDA-DM-98283 (Other: UT MD Anderson Cancer Center); NCI-G00-1742; CDR0000067734 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-04-06; First posted 2004-04-23 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage III multiple myeloma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute monoblastic leukemia and acute monocytic leukemia (M5); childhood acute monoblastic leukemia and acute monocytic leukemia (M5); T-cell large granular lymphocyte leukemia; B-cell chronic lymphocytic leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; L3 childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; non-T, non-B childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive childhood acute lymphoblastic leukemia; non-T, non-B, cALLa negative childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive, pre-B childhood acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; non-T, non-B adult acute lymphoblastic leukemia; non-T, non-B, cALLa positive adult acute lymphoblastic leukemia; non-T, non-B, cALLa positive, pre-B adult acute lymphoblastic leukemia; non-T, non-B, cALLa negative adult acute lymphoblastic leukemia; TdT positive adult acute lymphoblastic leukemia; TdT negative adult acute lymphoblastic leukemia; TdT negative childhood acute lymphoblastic leukemia; TdT positive childhood acute lymphoblastic leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute eosinophilic leukemia; childhood acute basophilic leukemia; childhood acute megakaryocytic leukemia (M7); untreated hairy cell leukemia; chronic myelomonocytic leukemia; acute undifferentiated leukemia; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute monocytic leukemia (M5b); previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); intraocular lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood large cell lymphoma; childhood large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Monocytic, Acute; Leukemia, Large Granular Lymphocytic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome | interventions — Cyclophosphamide; Ficusin; Methoxsalen; Thiotepa; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemo, RT + PSCT (Experimental): Chemotherapy, Radiation Therapy, and Peripheral Stem Cell Transplantation
  Interventions: Drug: Cyclophosphamide; Drug: Psoralen; Drug: Thiotepa; Procedure: Allogeneic bone marrow transplantation; Procedure: In vitro-treated peripheral blood stem cell transplantation (PBSCT); Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Cyclophosphamide — IV over 2 hours on days 2 and 3
  Other Names: Cytoxan; Neosar
Drug: Psoralen — Psoralen treated T-cell allogeneic transplant on day 9
  Other Names: Methoxsalen; 8-methoxypsoralen; UVADEX; Oxsoralen-Ultra; Oxsoralen; 8-MOP
Drug: Thiotepa — IV over 2 hours on day 1
Procedure: Allogeneic bone marrow transplantation — Preserved stem cell or bone marrow allogeneic transplant plus psoralen treated T-cell allogeneic transplant on day 9
Procedure: In vitro-treated peripheral blood stem cell transplantation (PBSCT) — Preserved stem cell or bone marrow allogeneic transplant plus psoralen treated T-cell allogeneic transplant on day 9
  Other Names: PBSCT
Radiation: Radiation Therapy (RT) — Whole body radiotherapy on days 5-8.
  Other Names: Radiotherapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by the chemotherapy or radiation therapy used to kill tumor cells. Sometimes the transplanted cells are rejected by the body's normal tissues. Transplanting donated cells that have been treated with psoralen may prevent this from happening.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy, radiation therapy, and psoralen-treated donor cells in treating patients who are undergoing peripheral stem cell transplantation for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of T-cells photochemically treated with psoralen and ultraviolet A given with peripheral stem cell transplantation in patients with hematologic malignancies or bone marrow failure myelodysplastic syndrome. II. Assess the toxicity of this treatment in these patients. III. Evaluate this regimen in terms of prevention of graft versus host disease and control of malignancy in these patients.

OUTLINE: This is a dose escalation, multicenter study of T-cells photochemically treated with psoralen and ultraviolet A. Patients receive thiotepa IV over 2 hours on day 1, cyclophosphamide IV over 2 hours on days 2 and 3, and whole body radiotherapy on days 5-8. Patients undergo preserved stem cell or bone marrow allogeneic transplant plus psoralen treated T-cell allogeneic transplant on day 9. Cohorts of 3-6 patients receive escalating doses of photochemically treated T-cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose limiting toxicities. Patients are followed for 100 days.

PROJECTED ACCRUAL: A maximum of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Hematologic malignancy, including acute myeloid or lymphoid leukemia of any FAB subtype, not in remission with chemotherapy or requiring bone marrow transplant OR Chronic myeloid leukemia, advanced beyond first chronic phase OR Myelodysplasia, including secondary to prior chemotherapy, with: Granulocyte count less than 500/mm3 OR Platelet count less than 50,000/mm3 OR High risk cytogenetic abnormalities such as +8, -7, -5, or 11q23 OR Intermediate or high grade lymphoma without response to initial therapy or in relapse OR Multiple myeloma without response to initial therapy or in relapse OR Stage IV low grade lymphoma or chronic lymphocytic leukemia not achieving remission with 2 regimens No aplastic anemia Related haploidentical donor (1-3 HLA-A, B, and/or DR mismatch) for collection of stem cells and whole blood T-cells required

PATIENT CHARACTERISTICS: Age: 6 months to 49 years Performance status: ECOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 1.5 mg/dL SGPT less than 3 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL Cardiovascular: Left ventricular ejection fraction at least 45% No symptoms or active treatment of left ventricular failure Pulmonary: Corrected DLCO at least 50% Other: No acute viral, bacterial, or fungal infection No prior transfusion associated graft versus host disease No other medical condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior immunotherapy or interferon alfa and recovered No prior autologous or allogeneic progenitor cell transplant Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 1999-05-28 (Actual); Primary Completion 2002-08-28 (Actual); Study Completion 2002-08-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of T-cells photochemically treated with psoralen and ultraviolet A | 100 days
  MTD defined as dose preceding that at which at least 2 of 3 patients experience dose limiting toxicities. Patients followed for 100 days.

CONTACTS AND LOCATIONS:
Overall Officials: James Gajewski, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org